CLINICAL TRIAL: NCT01476267
Title: An Open Label, Single Centre Study to Investigate the Metabolic Profile of Dalcetrapib After a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study of the Metabolic Profile of Dalcetrapib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WP27937
Record Dates: First submitted 2011-11-11; First posted 2011-11-22 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — dalcetrapib

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: dalcetrapib

INTERVENTIONS:
Drug: dalcetrapib — Single oral radiolabeled dose

SUMMARY:
This single center, open-label, non-randomized, one-treatment, one-period study will evaluate the metabolic profile and the safety of a single oral radiolabeled dose of dalcetrapib in male healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 45 to 65 years of age inclusive
* Body mass index (BMI) between 18 and 32 kg/m2 inclusive

Exclusion Criteria:

* Any concomitant disease or ongoing condition that in the investigator's opinion could interfere with the study or could pose an unacceptable risk to the subject
* Clinically significant abnormal laboratory values
* Infrequent bowel movements (e.g. less than one movement per 24 h on average)
* An intent to father children within 3 months of dosing
* Any external or internal radiotherapy with open (nuclear medicine) or sealed sources (brachy therapy)
* External irradiation (radiological examination) or internal radiation (diagnostic nuclear medicine procedure) within one year before study drug dosing; dental radiography and plain X-rays of the extremities are allowed before dosing

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (4.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Profile: Percentage of Free Thiophenol M1 in the Blood Plasma
Time Frame: up to Day 5
Measure: Mean (Standard Deviation); unit: Percentage of Free Thiophenol M1
Arm/Group | Single Arm
Number analyzed (Participants) | 6
Percentage of Free Thiophenol M1 | 37.5 (1.4)

2. Secondary Outcome: Correlation of Metabolic Profile With Enzyme/Transporter Genotypes
Time Frame: approximately 3 months
Population: Data was not collected
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=6)
Diarrhea (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No